CLINICAL TRIAL: NCT04601740
Title: A Multi-centre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Use of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in The Netherlands
Brief Title: A Research Study Looking at How Oral Semaglutide Works in People With Type 2 Diabetes in The Netherlands, as Part of Local Clinical Practice
Acronym: PIONEER REAL
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4643; U1111-1240-4249 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment.
  Interventions: Drug: Oral Semaglutide

INTERVENTIONS:
Drug: Oral Semaglutide — Patients will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.

SUMMARY:
The purpose of the study is to collect information on how Rybelsus® works in people with type 2 diabetes and to see if Rybelsus® can lower their blood sugar levels. Participants will get Rybelsus® as prescribed to them by the study doctor. The study will last for about 8-10 months. Participants will be asked to complete a questionnaire about how they take their Rybelsus® tablets. Participants will complete this questionnaire during their normally scheduled visit with the study doctor.

Participants will be asked to complete some questionnaires about their diabetes treatment. Participants will complete these during their normally scheduled visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Diagnosed with type 2 diabetes mellitus
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Available HbA1c value less than or equal to 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit'(V1) if in line with local clinical practice
* Treatment naïve to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than or equal to 14 days

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Treatment with any investigational drug within 30 days prior to enrolment into the study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Glycated haemoglobin (HbA1c ) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percent-points

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percent
Absolute change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Kilogram (Kg)
HbA1c <7% (Yes/No) | End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving the target value
HbA1c reduction >=1%-points and body weight reduction of >=5% (Yes/No) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving the reduction
HbA1c reduction >=1%-points and body weight reduction of >=3% (Yes/No) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving the reduction
Diabetes Treatment Satisfaction Questionnaire, change (DTSQc), relative treatment satisfaction | End of Study visit (V3) (week 34-44)
  Total score
Diabetes Treatment Satisfaction Questionnaire, status (DTSQs), change in absolute treatment satisfaction | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Total score

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Master Centre Netherlands, Alphen aan den Rijn, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Rudofsky G, Amadid H, Braae UC, Catrina SB, Kick A, Mandavya K, Roslind K, Saravanan P, van Houtum W, Jain AB. Oral Semaglutide Use in Type 2 Diabetes: A Pooled Analysis of Clinical and Patient-Reported Outcomes from Seven PIONEER REAL Prospective Real-World Studies. Diabetes Ther. 2025 Jan;16(1):73-87. doi: 10.1007/s13300-024-01668-6. Epub 2024 Nov 13. PMID 39535683
- [Derived] van Houtum W, Schrombges P, Amadid H, van Bon AC, Braae UC, Hoogstraten C, Herrings H. Real-World Use of Oral Semaglutide in Adults with Type 2 Diabetes in the PIONEER REAL Netherlands Multicentre, Prospective, Observational Study. Diabetes Ther. 2024 Aug;15(8):1749-1768. doi: 10.1007/s13300-024-01588-5. Epub 2024 Jun 11. PMID 38861137